CLINICAL TRIAL: NCT03763591
Title: Psychological Skills Group for Youth of Refugee and Immigrant Backgrounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jeffrey Winer, Research Fellow, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-P00029550
Record Dates: First submitted 2018-11-28; First posted 2018-12-04 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Stress, Psychological; Acculturation Problem
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychological Skills Group (e.g., Active Intervention) (Experimental): 10-week Psychological Skills Group.
  Interventions: Behavioral: Trauma Systems Therapy for Refugees Group Intervention

INTERVENTIONS:
Behavioral: Trauma Systems Therapy for Refugees Group Intervention — Psychological skills group for youth of refugee and immigrant backgrounds.

SUMMARY:
There are currently 28 million child refugees worldwide - approximately 1 in every 200 children on earth. To date, nearly one million forcibly displaced child migrants have been resettled in the United States. It is well documented that refugee and immigrant youth, especially forcibly displaced ethnic and cultural minority youth, present with alarmingly high rates of stress-related psychiatric illness (e.g., PTSD, depression, anxiety) and are grossly underserved by current mental health, medical, and social services. Previous research found that in a sample of 144 Somali refugee children resettled in the United States, only 8% of those who met full clinical criteria for PTSD received any mental health services. Through a process of community-based participatory research with refugee and immigrant communities and stake-holders the investigators have developed a multi-tiered psychological and systems intervention for refugee youth and families, Trauma Systems Therapy for Refugees (TST-R), that includes community outreach and advocacy, group psychological treatment, office-based psychotherapy, and home-based services.

Whereas TST-R is one of the only empirically-based behavioral health treatment models for refugee youth, it has only been studied as a full intervention model; financial and staffing resource barriers have limited the wide-spread adoption of the model. This obstacle noted, implementing one high-impact component of this multi-tier intervention (i.e., protocol-driven group treatments) may provide significant benefit while also being easily scalable. Implementing time-limited (i.e., 10 week) manual-based group psychological interventions focused on culturally-responsive strategies to support refugee youth with, and at-risk for, PTSD, depression, and anxiety, may be an efficient and cost effective means of (1) reducing psychiatric symptoms for refugee and migrant youth with present symptoms, (2) preventing symptom onset for those at risk, and (3) enhancing cultural identity self-concept, subjective social belongingness, and psychological resilience (e.g., ability to thrive in the context of adversity). Furthermore, if effective, treatment groups can importantly function as a destigmatizing treatment gateway and triage to other services for youth who require a higher level of care (e.g., individual psychotherapy and medication management).

ELIGIBILITY:
Inclusion Criteria:

* Age 15-18 years old living in the Greater Boston Area.
* Of refugee or immigrant background (e.g., youth or a parent arrived to the USA as a refugee or immigrant)
* No current plans to move from Greater Boston Area within the next 6 months
* Conversationally proficient in English language

Exclusion Criteria:

* Not able to attend group once a week for 10 weeks
* Medical, cognitive, or other health or psychosocial issue that would prevent consistent and engagement and participation in group.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Depression Symptoms | Change from Baseline after 10 weeks of the intervention.
  Depression as measured by the Patient Health Questionnaire-9 (PHQ-9). Self-report depression scale, higher scores mean greater symptoms of depression (e.g., worse outcome). Total score sum may range from 0 to 27.
Anxiety Symptoms | Change from Baseline after 10 weeks of the intervention.
  Anxiety as measured by the Generalized Anxiety Disorder-7 (GAD-7). Self-report anxiety scale, higher scores mean greater symptoms of anxiety (e.g., worse outcome). Total score sum may range from 0 to 21.
Post Traumatic Stress Disorder (PTSD) Symptoms | Change from Baseline after 10 weeks of the intervention.
  PTSD as measured by the STRESS (Structured Trauma-Related Experiences and Symptoms Screener). Self-report PTSD scale, higher scores mean greater symptoms of PTSD (e.g., worse outcome). Total score sum may range from 0 to 68.
Cultural Identity Self-Concept | Change from Baseline after 10 weeks of intervention.
  Cultural Identity Self-Concept measured with social and cultural identities adapted version of Cognitive Fusion Questionnaire (CFQ). Self-report measure. Higher scores indicate greater cognitive and emotional suffering related to social and cultural identity self-concept (example item: "my thoughts about my social and cultural identities cause me distress or emotional pain." Total score sum may range from 0 to 42. Higher scores indicate worse outcome.
Self-Efficacy | Change from Baseline after 10 weeks of intervention.
  Self-Efficacy measured by New General Self-Efficacy Scale (NGSES). Self-report measure. Higher scores indicate greater perceived ability to accomplish goals and overcome challenges (example item: "I will be able to achieve most of the goals that I have set for myself.") Total score sum may range from 0 to 48. Higher scores indicate better outcome.
Social Belongingness | Change from Baseline after 10 weeks of intervention.
  Social Belongingness as measured by the General Belongingness Scale (GBS). Self-report measure. Higher scores indicate greater sense of social belongingness (example item: "I feel connected with others.") Total score sum may range from 0 to 72. Higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellis BH, Miller AB, Abdi S, Barrett C, Blood EA, Betancourt TS. Multi-tier mental health program for refugee youth. J Consult Clin Psychol. 2013 Feb;81(1):129-40. doi: 10.1037/a0029844. Epub 2012 Aug 27. PMID 22924331
- [Background] Ellis BH, MacDonald HZ, Lincoln AK, Cabral HJ. Mental health of Somali adolescent refugees: the role of trauma, stress, and perceived discrimination. J Consult Clin Psychol. 2008 Apr;76(2):184-93. doi: 10.1037/0022-006X.76.2.184. PMID 18377116
- [Background] Bogic M, Njoku A, Priebe S. Long-term mental health of war-refugees: a systematic literature review. BMC Int Health Hum Rights. 2015 Oct 28;15:29. doi: 10.1186/s12914-015-0064-9. PMID 26510473
- [Background] Grasso DJ, Felton JW, Reid-Quinones K. The Structured Trauma-Related Experiences and Symptoms Screener (STRESS): Development and Preliminary Psychometrics. Child Maltreat. 2015 Aug;20(3):214-20. doi: 10.1177/1077559515588131. Epub 2015 Jun 19. PMID 26092442
- [Background] Lustig SL, Kia-Keating M, Knight WG, Geltman P, Ellis H, Kinzie JD, Keane T, Saxe GN. Review of child and adolescent refugee mental health. J Am Acad Child Adolesc Psychiatry. 2004 Jan;43(1):24-36. doi: 10.1097/00004583-200401000-00012. PMID 14691358
- [Background] Alegria M, Vallas M, Pumariega AJ. Racial and ethnic disparities in pediatric mental health. Child Adolesc Psychiatr Clin N Am. 2010 Oct;19(4):759-74. doi: 10.1016/j.chc.2010.07.001. PMID 21056345
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Gillanders DT, Bolderston H, Bond FW, Dempster M, Flaxman PE, Campbell L, Kerr S, Tansey L, Noel P, Ferenbach C, Masley S, Roach L, Lloyd J, May L, Clarke S, Remington B. The development and initial validation of the cognitive fusion questionnaire. Behav Ther. 2014 Jan;45(1):83-101. doi: 10.1016/j.beth.2013.09.001. Epub 2013 Sep 18. PMID 24411117
- [Background] Malone, G. P., Pillow, D. R., Osman, A. (2012). The General Belongingness Scale (GBS): Assessing achieved belongingness. Personality and Individual Differences, 52(3), 311-316.
- [Background] Chen, G., Gully, S. M., & Eden, D. (2001). Validation of a New General Self-Efficacy Scale. Organizational Research Methods, 4(1), 62-83.